CLINICAL TRIAL: NCT00817583
Title: Phse II Study of Induction Chemotherapy With TPF Regimen Followed by Concurrent Chemoradiotherapy for Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Chemotherapy Followed by Concurrent Chemoradiotherapy for Nasopharyngeal Carcinoma (NPC)
Acronym: TPF for NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: cancer hospital, Fudan University, cancer hospital, Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC20081; NPC20081; NPC20081-1
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Phase 2 Clinical Trial; NPC; neoadjuvant chemotherapy; concurrent chemoradiation
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; Cisplatin; Fluorouracil; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All patients will receive docetaxel 75 mg/m2 on day 1; cisplatin 75 mg/m2 on day 1; and a continuous intravenous fluorouracil infusion at 500 mg/m2/d on days 1 through 5. Cycles are repeated every 21 days for a total of two cycles. Patients then will receive definitive radiotherapy with 3D-CRT or IMRT, and cisplatin (40mg/m2) weekly during external radiotherapy.The radiation dose is 66-76Gy to the GTV, 60Gy to CTV1, and 54Gy to CTV2.
  Interventions: Drug: docetaxel, cisplatin, fluorouracil; Radiation: 3D-CRT (three-dimensional conformal radiation therapy) or IMRT (intensity-modulated radiation therapy)

INTERVENTIONS:
Drug: docetaxel, cisplatin, fluorouracil — neoadjuvant chemotherapy:docetaxel 75 mg/m2 on day 1; cisplatin 75 mg/m2 on day 1; continuous fluorouracil infusion at 500 mg/m2/d on days 1 through 5.
  concurrent chemotherapy:cisplatin 40 mg/m2 weekly
Radiation: 3D-CRT (three-dimensional conformal radiation therapy) or IMRT (intensity-modulated radiation therapy)

SUMMARY:
The primary objective of this study is to determine the response rate, tolerance and overall survival in patients with stage III, IVa, IVb NPC treated with neoadjuvant chemotherapy (TPF regimen) and concurrent chemoradiation.

Secondary objectives of the study are to evaluate the distant metastases free survival, and disease-free survival of patients with stage III,IVa, IVb NPC treated with this regimen.

The third objective of this study is to evaluate who may benifit from this treatment regimen.

DETAILED DESCRIPTION:
Concurrent chemoradiation is the standard treatment for locally advanced NPC. The survival benefit gained from adding induction chemotherapy to concurrent chemoradiation has not been defined yet. In the present clinical study, we hope to assess the tolerance and survival benefits of induction chemotherapy followed by concurrent chemoradiation in patients with stage III, IVa and IVb NPC.

ELIGIBILITY:
Inclusion Criteria:

* -Histopathologically proved WHO type II and type III carcinoma of the nasopharynx.
* Stage Ⅲ, IVa and IVb disease
* KPS >70
* Age between 18-70
* Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count (AGC) of > 2000 cells/mm3, platelet count of > 100,000 cells/mm3 (pre treatment without intervention). Bilirubin < 1.5 mg/dl, AST or ALT<2 x upper normal, serum creatinine<1.5mg/dl, creatinine clearance >50ml/min.
* the primary tumor or involved lymph node must be more than 2CM in diameter.
* No prior radiation treatment to the head and neck or any prior chemotherapy
* Patients with no prior malignancy (not include basal cell carcinoma of skin)

Exclusion Criteria:

* Evidence of metastases (below the clavicle or distant) by clinical or radiographic examinations.
* Prior radiotherapy to the head and neck region for any reason.
* Initial surgical treatment excluding diagnostic biopsy of the primary site or neck disease.
* Patients with previous or simultaneous primaries, excluding basal cell carcinoma or squamous cell carcinoma of skin.
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 and 5 years

SECONDARY OUTCOMES:
distant metastases free survival , and disease-free survival | 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: XiaoShen WANG, M.D., Principal Investigator — Department of Radiation Oncology, Cancer Hospital, Fudan University; ChaoSu HU, M.D., Study Chair — Department of Radiation Oncology, Cancer Hospital, Fudan University; ChunYing Shen, M.D., Principal Investigator — Department of Radiation Oncology, Cancer Hospital, Fudan University; HongMei Ying, M.D., Principal Investigator — Department of Radiation Oncology, Cancer Hospital, Fudan University
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality, China